CLINICAL TRIAL: NCT04609202
Title: Measuring the Effect of Person Centered, Nurse Led Care on Health-related Quality of Life in Patients With Atrial Fibrillation
Brief Title: Person Centered Nurse Led Atrial Fibrillation Care
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Umeå University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Flimmerstudie2020
Record Dates: First submitted 2020-10-09; First posted 2020-10-30 (Actual); Last update posted 2025-04-02 (Actual); Status verified 2025-03

CONDITIONS: Atrial Fibrillation
Keywords: atrial fibrillation; person centred care; health related quality of life; nurse led
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Nurse led person centred care (Experimental): Participants in the nurse led, person centred care arm will receive person centred follow up after hospitalization for atrial fibrillation. The person centred care and usual care routines are provided by nurses.
  Interventions: Behavioral: Nurse led person centred care
- Usual care (Active Comparator): Participants in the usual care arm will receive care as usual, ie follow up by doctors after hospitalization for atrial fibrillation.
  Interventions: Other: Usual care

INTERVENTIONS:
Behavioral: Nurse led person centred care — Person centred care include patiens narratives, partnership and documentation of a health plan.
  Arms: Nurse led person centred care
Other: Usual care — Usual care provided by doctors
  Arms: Usual care

SUMMARY:
The aim of the study is to evaluate the effect of a person-centred nurse-led outpatient clinic on health related quality of life, for persons with AF. Secondary outcomes are effects on anxiety, depression, illness perception, symtom burden, life style and health economics.

DETAILED DESCRIPTION:
The aim of the study is to evaluate the effect of a person-centred nurse-led outpatient clinic on health related quality of life, for persons with AF. Secondary outcomes are effects on anxiety, depression, illness perception, symtom burden, life style and health economics.

We plan a randomized controlled trial comparing person centred nurse led care vs. standard care. A sample size of 100 persons per group will be recruited.

Data will be collected through questionnaires, medical records, interviews.

ELIGIBILITY:
Inclusion Criteria:

* patients aged > 18 years with diagnosis of atrial fibrillation, referred for follow up after atrial fibrillation, able to provide informed consent and able and willing to fill in questionnaires.

Exclusion Criteria:

* Atrial flutter diagnosis, Severe heart failure (corresponding to NYHA IIIB and NYHA IV), Cardiac surgery < 3 month prior to hospitalization for atrial fibrillation, planned surgical procedures (catheter ablation, cardiac surgery), Atrial fibrillation in connection with acute coronary syndrome or infection, not able to fill in questionnaires.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2020-10-19 (Actual); Primary Completion 2025-07-10 (Estimated); Study Completion 2025-07-10 (Estimated)

PRIMARY OUTCOMES:
Health related quality of life measured by EuroQol-5D (EQ-5D) questionnaire | Baseline, 6 month and 1 year
  Change from baseline in health related quality of life, measured by EuroQol-5D (EQ-5D) questionnaire at six month and one year. EQ-5D measure Health related quality of life with scores (5 items) and a scale (0-100).
Arrhythmia related quality of life measured by Arrhythmia-Specific questionnaire in Tachycardia and Arrhythmias (ASTA) | Baseline, 6 month and 1 year
  Change from baseline in arrhythmia related quality of life, measured by Arrhythmia-Specific questionnaire in Tachycardia and Arrhythmias (ASTA), at six month and one year. ASTA is a validated questionnaire with a 13-item arrhythmia related quality of life scale. The scores for the total scale range between 0 and 39, with higher scores reflecting more negative effects on HRQoL.

SECONDARY OUTCOMES:
Anxiety measured by Hospital Anxiety and Depression Scale (HADS) | Baseline, 6 month and 1 year
  Change from baseline in anxiety, measured by Hospital Anxiety and Depression Scale (HADS) at six month and one year. HADS-anxiety ranges from 0 to 21; higher scores indicate higher anxiety complains.
Depression measured by Hospital Anxiety and Depression Scale (HADS) | Baseline, 6 month and 1 year
  Change from baseline in depression, measured by Hospital Anxiety and Depression Scale (HADS), at six month and one year. HADS-depression ranges from 0 to 21; higher scores indicate higher depression complains.
Symptom burden measured by Arrhythmia-Specific questionnaire in Tachycardia and Arrhythmias (ASTA) | Baseline, 6 month and 1 year
  Change from baseline in symptom burden, measured by Arrhythmia-Specific questionnaire in Tachycardia and Arrhythmias (ASTA), at six month and one year. ASTA is a validated questionnaire with a 9-item symptom scale, each with a score of 0-4, The scores for the total scale range between 0 and 27, with higher scores reflecting higher symptom burden.
Lifestyle habits-smoking, measured by questionnaire, | Baseline, 6 month and 1 year
  Change from baseline in lifestyle habits-smoking, measured by questionnaire (developed by The Swedish National Board of Health and Welfare), whether the patient is non smoker, prior smoker or current smoker (self-report), at six month and one year.
Lifestyle habits-diet by questionnaire | Baseline, 6 month and 1 year
  Change from baseline in lifestyle habits-diet, measured by a questionnaire (developed by The Swedish National Board of Health and Welfare) with 5 items about eating habits, at six month and one year.
Lifestyle habits-physical activity by questionnaire | Baseline, 6 month and 1 year
  Change from baseline in lifestyle habits-physical activity, measured by a questionnaire (developed by The Swedish National Board of Health and Welfare) with 2 items about physical activity habits, at six month and one year.
Lifestyle habits-alcohol use by questionnaire | Baseline, 6 month and 1 year
  Change from baseline in lifestyle habits-alcohol use, measured by a questionnaire (developed by The Swedish National Board of Health and Welfare) with 3 items about alcohol use, at six month and one year.
Illness perception measured by Brief Illness Perception Questionnaire (B-IPQ) | Baseline, 6 month and 1 year
  Change from baseline in illness perception, measured by Brief Illness Perception Questionnaire (B-IPQ) at six month and one year. B-IPQ measures illness perception and is a 9-item validated questionnaire. 8 items are scored 0-10, the 9th item is a question of cause and answering in text.
Quality-adjusted life years,(QALYs) gathered with EuroQol-5D (EQ-5D) questionnaire. | Baseline to 1 year
  Change from baseline in quality-adjusted life years (QALYs) at one year. The EuroQoL-5D-3L (EQ-5D) will be used for the quality of life dimension, while the time elapsed between each EQ-5D measurement will be considered for the time dimension.

CONTACTS AND LOCATIONS:
Overall Officials: Karin H Ängerud, Principal Investigator — Umeå University
Locations (1):
- Norrlands Universitetssjukhus, Umeå, Region Västerbotten, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Holmlund L, Hornsten C, Valham F, Olsson K, Hornsten A, Katsoularis I, Salonen L, Angerud KH. The effects of a nurse-led, person-centred outpatient clinic on patient-reported outcomes in patients with atrial fibrillation - a randomised controlled trial. Eur J Cardiovasc Nurs. 2026 Jan 29:zvag028. doi: 10.1093/eurjcn/zvag028. Online ahead of print. PMID 41610156